CLINICAL TRIAL: NCT03274531
Title: Pharmacists Intervention to Improve Hypertension Management in Primary Care (APOTHECARE): A Cluster-randomized Trial
Brief Title: Pharmacists Intervention to Improve Hypertension Management in Primary Care
Acronym: APOTHECARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilhelminenspital Vienna (Other)
Collaborators: Österreichische Apothekerkammer, Landesgeschäftsstelle Niederösterreich (Unknown); Association for the Promotion of Research in Atherosclerosis, Thrombosis and Vascular Biology (Other); Institute for Cardiometabolic Diseases, Karl Landsteiner Society (Unknown)
Responsible Party: Principal Investigator, Miklos Rohla, MD, Wilhelminenspital Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APOTHECARE
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective, cluster randomized, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Immediate referral of hypertensive patients to the attending physician based on automated office blood pressure measurements
  Interventions: Behavioral: Referral of hypertensive patients to the attending physician
- Observational Arm (No Intervention): Repeated automated office blood pressure measurements and referral of hypertensive patients to the attending physician after completion of the trial

INTERVENTIONS:
Behavioral: Referral of hypertensive patients to the attending physician — Immediate referral to the treating physician in case of elevated automated office blood pressure measurements
  Arms: Interventional Arm

SUMMARY:
Arterial hypertension is the single largest contributor to mortality world-wide, and only 30-50% of diagnosed and treated patients achieve their blood pressure goal. The APOTHECARE trial is designed to identify treated patients with uncontrolled hypertension in community pharmacies in order to improve blood pressure control through intensification of antihypertensive therapy.

DETAILED DESCRIPTION:
Patients with medically treated arterial hypertension, who attend a pharmacy in order to obtain their antihypertensive medication are invited to participate in the trial.

The main inclusion criteria is uncontrolled hypertension, as determined by an automated office blood pressure measurement at a threshold of 135/85 mmHg.

Main exclusion criteria include a first-ever prescription of an antihypertensive agent, resistant hypertension, systolic blood pressure ≥ 180 mmHg and dialysis.

Randomization occurs on the level of pharmacies (cluster randomization).

Patients in the interventional arm are immediately referred to their treating physician for up-titration of antihypertensive therapy. Re-examination of automated automated office blood-pressure occurs in the respective pharmacy, and patients are referred to their treating physician again if required. These measures are accompanied by a structured and educational blood pressure record card.

Patients in the observational arm undergo periodic automated office blood pressure measurements and are referred to their treating physician at the end of the trial in case of persistently uncontrolled blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Medically pre-treated arterial hypertension
* Automated office blood pressure ≥ 135 mmHg systolic or ≥ 85 mmHg diastolic

Exclusion Criteria:

* First ever prescription of antihypertensive medication
* First prescription of a new antihypertensive substance or dose adjustment
* Prior therapy with 4 or more different antihypertensive substances
* Systolic blood pressure ≥ 180 mmHg
* Dialysis
* Adherence to the study protocol not to be anticipated
* Inclusion into the study at another study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with systolic blood pressure <135 mmHg and diastolic blood pressure < 85 mmHg at 10 weeks of follow-up (automated office blood pressure measurement) | 10 weeks
  Primary endpoint

SECONDARY OUTCOMES:
Change in average systolic blood pressure (automated office blood pressure measurement) | 10 weeks
  Secondary endpoint
Change in average systolic blood pressure (automated office blood pressure measurement) | 20 weeks
  Secondary endpoint
Proportion of patients with systolic blood pressure <135 mmHg and diastolic blood pressure < 85 mmHg (automated office blood pressure measurement) | 20 weeks
  Secondary endpoint
Proportion of patients with systolic blood pressure <135 mmHg and diastolic blood pressure < 85 mmHg (home blood pressure, mean of available readings) | 20 weeks
  Secondary endpoint, patients with available home blood pressure measurements

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Rohla, MD, Principal Investigator — 3rd Medical Department, Cardiology and Intensive Care Medicine, Wilhelminenhospital, Vienna, Austria; Thomas W Weiss, MD, PhD, Study Chair — 3rd Medical Department, Cardiology and Intensive Care Medicine, Wilhelminenhospital, Vienna, Austria
Locations (54):
- Austria (54):
  - Buchen-Apotheke, Alland
  - Apotheke Bad Erlach, Bad Erlach
  - Kur-Apotheke, Bad Vöslau
  - Landschafts-Apotheke, Baden
  - Apotheke Am Goettweiger, Furth
  - Oetscherland-Apotheke, Gaming
  - Apotheke zum heiligen Georg, Gaweinstal
  - Apotheke Gmuend Neustadt, Gmünd
  - Apotheke Zum Auge Gottes, Gmünd
  - Marien-Apotheke, Gramatneusiedl
  - St. Georgs-Apotheke, Himberg
  - Apotheke Zu Maria Trost, Kirchberg am Wagram
  - Stadt-Apotheke, Klosterneuburg
  - Die Blaue Apotheke, Klosterneuburg
  - Kreis-Apotheke Zum schwarzen Adler, Korneuburg
  - Adler-Apotheke, Langenlois
  - Kamptal-Apotheke, Langenlois
  - Kronen-Apotheke, Lilienfeld
  - Apotheke Zur Madonna, Neunkirchen
  - Merkur-Apotheke, Neunkirchen
  - Triesting-Apotheke,, Oberwaltersdorf
  - Apotheke Zum heiligen Georg, Pitten
  - Apotheke Zum St. Nikolaus, Pottendorf
  - Apotheke Zur Mariahilf, Pöggstall
  - Apotheke Purgstall, Purgstall
  - Wallhof-Apotheke, Rannersdorf
  - Apotheke Sued, Sankt Pölten
  - Center Apotheke, Sankt Pölten
  - Hippolyt-Apotheke, Sankt Pölten
  - Rosen-Apotheke, Sankt Pölten
  - Stadt-Apotheke, Schrems
  - Linden-Apotheke, Seitenstetten Markt
  - Johannes-Apotheke, Traisen
  - Apotheke Zur Mutter Gottes, Traismauer
  - Activ Apotheke Tribuswinkel, Tribuswinkel
  - Urania Apotheke, Vienna
  - Siebenbrunnen Apotheke, Vienna
  - Heilfried Apotheke, Vienna
  - Ludwigs Apotheke, Vienna
  - Friedrichs Apotheke, Vienna
  - Linden Apotheke, Vienna
  - Adler Apotheke, Vienna
  - Arkaden Apotheke, Vienna
  - Rosen Apotheke, Vienna
  - Apotheke Neu Kagran, Vienna
  - St. Hubertus Apotheke, Vienna
  - Birken Apotheke, Vienna
  - Apotheke Zur Mariahilf, Wiener Neustadt
  - Bahnhof-Apotheke, Wiener Neustadt
  - Zehnerguertel-Apotheke, Wiener Neustadt
  - Apotheke Wimpassing, Wimpassing
  - Apotheke Zur heiligen Dreifaltigkeit, Wolkersdorf
  - Apotheke Zum schwarzen Adler, Zwettl Stadt
  - Kuenringer Apotheke, Zwettl Stadt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohla M, Haberfeld H, Tscharre M, Huber K, Weiss TW. Pharmacist interventions to improve blood pressure control in primary care: a cluster randomised trial. Int J Clin Pharm. 2023 Feb;45(1):126-136. doi: 10.1007/s11096-022-01452-1. Epub 2022 Nov 8. PMID 36346543